CLINICAL TRIAL: NCT00003593
Title: Treatment of Children With Down Syndrome (DS) and Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), and Transient Myeloproliferative Disorder (TMD): A Phase III Group-Wide Study
Brief Title: Chemotherapy in Treating Children With Down Syndrome and Myeloproliferative Disorder, Acute Myelogenous Leukemia, or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2971; COG-A2971 (Other: Children's Oncology Group); CCG-A2971 (Other: Children's Cancer Group); POG-A2971 (Other: Pediatric Oncology Group); CCG-29701 (Other: Children's Cancer Group); CDR0000066664 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: childhood myelodysplastic syndromes; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; de novo myelodysplastic syndromes; childhood acute minimally differentiated myeloid leukemia (M0); childhood acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); myelodysplastic/myeloproliferative neoplasm, unclassifiable; juvenile myelomonocytic leukemia; chronic myelomonocytic leukemia; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myelomonocytic, Chronic | interventions — Asparaginase; Cytarabine; Daunorubicin; Methotrexate; Hydrocortisone; hydrocortisone hemisuccinate; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: TMD patients only (Experimental): Patients are observed if their transient myeloproliferative disorder (TMD) does not require intervention. Patients who require therapy for TMD undergo leukapheresis or exchange transfusion for up to 3 consecutive days. If the TMD does not resolve or there is significant organ involvement, patients receive low-dose cytarabine IV continuously on days 0-4. Treatment repeats at least every 2 weeks for up to 4 courses. Patients who experience a recurrence of TMD at least 8 weeks after resolution or have refractory disease may proceed to group II for further treatment. patients will continue to be followed for remission induction, EFS, DFS and OS regardless of the type of leukemia that develops.
  Interventions: Drug: cytarabine
- Arm B: AML/MDS patients only (Experimental): (closed to accrual as of 6/24/04 except for patients first enrolled in group I): Patients receive induction therapy comprising cytarabine IV continuously, daunorubicin hydrochloride IV continuously, and oral thioguanine twice daily on days 0-3. Treatment repeats every 28 days for 4 courses. Patients with no CNS disease at diagnosis receive cytarabine intrathecally (IT) on day 0. Patients with CNS disease at diagnosis receive cytarabine IT on days 0, 5, and 7. If CNS disease persists on day 7, patients receive up to 6 courses of cytarabine IT, therapeutic hydrocortisone IT, and methotrexate IT, twice weekly beginning on day 10. Asparaginase during Intensification 1 day 1 hour 18.
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: methotrexate; Drug: therapeutic hydrocortisone; Drug: thioguanine

INTERVENTIONS:
Drug: asparaginase — Given IV
  Other Names: Elspar; Kidrolase; Crasnitin; Leunase; NSC #109229
  Arms: Arm B: AML/MDS patients only
Drug: cytarabine — Given IT
  Other Names: cytosine arabinoside; AraC; Cytosar; NSC #063878
Drug: daunorubicin hydrochloride — Given IV
  Other Names: daunomycin; DNR; Cerubidine; NSC #82151
  Arms: Arm B: AML/MDS patients only
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; NSC #000740
  Arms: Arm B: AML/MDS patients only
Drug: therapeutic hydrocortisone — Given IT
  Other Names: Cortef; Solu-cortef; NSC #010483
  Arms: Arm B: AML/MDS patients only
Drug: thioguanine — Given IV
  Other Names: 6-thioguanine; 6-TG; NSC # 000752
  Arms: Arm B: AML/MDS patients only

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase III trial to study the effectiveness of combination chemotherapy in treating children who have Down syndrome and myeloproliferative disorder, acute myelogenous leukemia, or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of reduced-dose induction and intensification chemotherapy, in terms of remission rate, disease-free survival rate, and acute morbidity and mortality, in children with Down syndrome and acute myelogenous leukemia or myelodysplastic syndromes.
* Define the understanding of the natural history of transient myeloproliferative disorder (TMD) in children with Down syndrome.
* Determine whether there is a reduction of sequelae in long-term survivors after treatment with this regimen.
* Determine the incidence of subsequent leukemia in patients with transient myeloproliferative disorder treated with this regimen.
* Determine the predictive risk factors for developing subsequent leukemia in patients with transient myeloproliferative disorder treated with this regimen.

OUTLINE: This is a multicenter study.

* Group I: Patients are observed if their transient myeloproliferative disorder (TMD) does not require intervention. Patients who require therapy for TMD undergo leukapheresis or exchange transfusion for up to 3 consecutive days. If the TMD does not resolve or there is significant organ involvement, patients receive low-dose cytarabine IV continuously on days 0-4. Treatment repeats at least every 2 weeks for up to 4 courses. Patients who experience a recurrence of TMD at least 8 weeks after resolution or have refractory disease may proceed to group II for further treatment.
* Group II (closed to accrual as of 6/24/04 except for patients first enrolled in group I): Patients receive induction therapy comprising cytarabine IV continuously, daunorubicin IV continuously, and oral thioguanine twice daily on days 0-3. Treatment repeats every 28 days for 4 courses. Patients with no CNS disease at diagnosis receive cytarabine intrathecally (IT) on day 0. Patients with CNS disease at diagnosis receive cytarabine IT on days 0, 5, and 7. If CNS disease persists on day 7, patients receive up to 6 courses of cytarabine IT, hydrocortisone IT, and methotrexate IT, twice weekly beginning on day 10.

Patients who achieve remission after induction therapy receive 2 courses of intensification therapy, for approximately 4 months. During the first course, patients receive cytarabine IV over 3 hours twice daily on days 0, 1, 7, and 8. Patients also receive asparaginase intramuscularly on days 1 and 8. The second course of therapy comprises CNS prophylaxis. Patients with no CNS disease at diagnosis or whose CNS disease resolved by day 7 of induction therapy receive cytarabine IT on days 0, 7, and 14. Patients with persistent CNS disease on day 7 of induction therapy receive cytarabine IT, hydrocortisone IT, and methotrexate IT on days 0, 7, and 14.

Patients are followed monthly for 18 months, every 3 months for 1 year, every 6 months for 2.5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 70 patients with acute myeloid leukemia or myelodysplastic syndromes will be accrued for this study within 3.2 years. A total of 88 patients with transient myeloproliferative disorder who enter remission will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytogenetically proven Down Syndrome (constitutional trisomy 21) with transient myeloproliferative disorder (TMD), myelodysplastic syndromes (MDS), or acute myelogenous leukemia (AML)

  * Must be confirmed by bone marrow aspirate, cerebrospinal fluid exam, or blood test
  * Trisomy 21 mosaicism allowed
* Group I:

  * Diagnosis of TMD in patients no older than 90 days at initial presentation
  * Must have nonerythroid blasts (any amount) in the peripheral blood and one of the following:

    * Verification with a second sample
    * More than 5% bone marrow blasts
    * Hepatomegaly and/or splenomegaly
    * Lymphadenopathy
    * Cardiac or pleural effusions OR
  * Histologically or cytologically proven TMD with blasts in an affected organ or in fluid (pericardial, pleural, or peritoneal)
  * Bone marrow aspirate is required
* Group II (closed to accrual as of 6/24/04):

  * Diagnosis of MDS or AML (except M3 subtype) in patients older than 90 days with more than 29% blasts in bone marrow (with or without history of TMD), or any of the following histologies:

    * Refractory anemia (RA)
    * RA with excess blasts (RAEB)
    * RAEB in transformation
    * RA with ringed sideroblasts (RARS)
    * Primary cytopenia (later confirmed by bone marrow aspirate as due to marrow hypoplasia) defined by one or more of the following:

      * Absolute neutrophil count less than 500/mm^3
      * Untransfused platelet count less than 30,000/mm^3
      * Untransfused hemoglobin less than 8 g/dL
* The following diagnoses will be observed only:

  * RA with mild cytopenias*
  * RARS with mild cytopenias*
  * Mild primary cytopenias (one or more) without dysplasia (confirmed by hypoplastic bone marrow exam) NOTE: * Platelet count 30-150,000/mm3, absolute neutrophil count 500-1,499/mm3, and hemoglobin greater than 8 g/dL
* Granulocytic sarcoma (chloroma), with or without bone marrow involvement, allowed

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 21 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* See Disease Characteristics

Renal:

* Not specified

Cardiovascular:

* Shortening fraction greater than 27% by echocardiogram* OR
* Ejection fraction greater than 47% by radionuclide angiogram* NOTE: *For patients with MDS and AML (as of 2/24/04, previously diagnosed MDS or AML closed to accrual; MDS or AML that develops (secondary to TMD) after study enrollment or MDS that requires initial observation [with or without subsequent treatment] allowed)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy for TMD allowed
* No prior chemotherapy for malignancy

Endocrine therapy:

* Concurrent topical or inhaled steroids for other conditions allowed

Radiotherapy:

* No prior radiotherapy for malignancy

Surgery:

* Not specified

Other:

* No prior antileukemic therapy
* Prior enrollment on this study for TMD allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 254 (Actual)
Dates: Start 1999-06; Primary Completion 2007-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Gamis, MD, MPH, Study Chair — Children's Mercy Hospital Kansas City
Locations (237):
- United States (209):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish RiteCampus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital at University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Perentesis JP, Alonzo TA, Gerbing R, et al.: Polymorphism in folate metabolism and outcomes of therapy in children with AML with and without Down Syndrome. [Abstract] Blood 102 (11 Pt 1): A-479, 2003.
- [Result] Sorrell AD, Alonzo TA, Hilden JM, Gerbing RB, Loew TW, Hathaway L, Barnard D, Taub JW, Ravindranath Y, Smith FO, Arceci RJ, Woods WG, Gamis AS. Favorable survival maintained in children who have myeloid leukemia associated with Down syndrome using reduced-dose chemotherapy on Children's Oncology Group trial A2971: a report from the Children's Oncology Group. Cancer. 2012 Oct 1;118(19):4806-14. doi: 10.1002/cncr.27484. Epub 2012 Mar 5. PMID 22392565
- [Result] Gamis AS, Alonzo TA, Gerbing RB, Hilden JM, Sorrell AD, Sharma M, Loew TW, Arceci RJ, Barnard D, Doyle J, Massey G, Perentesis J, Ravindranath Y, Taub J, Smith FO. Natural history of transient myeloproliferative disorder clinically diagnosed in Down syndrome neonates: a report from the Children's Oncology Group Study A2971. Blood. 2011 Dec 22;118(26):6752-9; quiz 6996. doi: 10.1182/blood-2011-04-350017. Epub 2011 Aug 17. PMID 21849481
- [Result] Gamis AS, Alonzo TA, Hilden JM, et al.: Outcome of Down syndrome (DS) children with acute myeloid leukemia (AML) or myelodysplasia (MDS) treated with a uniform prospective clinical trial initial report of the COG trial A2971. [Abstract] Blood 108 (11): A-15, 2006.
- [Result] Sharma M, Alonzo TA, Sorrell A, et al.: Uniform approach better defines natural history of transient myeloproliferative disorder (TMD) in Down syndrome (DS) neonates: outcomes from Children's Oncology Group (COG) study A2971. [Abstract] Blood 108 (11): A-376, 2006.